CLINICAL TRIAL: NCT00550940
Title: Emotion/Behavior Problems, Neuropsychological Functioning, and Parental Adjustment in Children and Adolescents With Epilepsy
Brief Title: Emotion/Behavior Problems, Neuropsychological Functioning, and Parental Adjustment in Children With Epilepsy
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200705066R
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-04

CONDITIONS: Epilepsy
Keywords: epilepsy; attention; emotion; behavior problems; child; adolescent
MeSH Terms: conditions — Epilepsy; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to Investigate characteristics and prevalence of emotion/behavior problems in child and adolescents with epilepsy; to identify the associated factors and their effects on these children/adolescents; and to examine their attention by using Conners' Continuous Performance Test (CPT).

DETAILED DESCRIPTION:
Child and adolescents with epilepsy often have comorbid conditions such as emotion/behavior problems and attention deficit, which usually result in great impact on their individual functioning and their family. Neurological factors (e.g. central neural system disease, mental retardation, and epilepsy factors), demographic factors (low socioeconomic, age, gender), family factors, child's attitude to epilepsy, parental psychopathology and their attitude may associate with the presentation of behavior and attention in child and adolescents with epilepsy. In addition, these risk factors may affect via some pathways. Previous studies were conducted mainly in Caucasians, and few researches were conducted in Chinese population. Furthermore, previous studies demonstrated inconsistent findings regarding the related risk factors for epilepsy. Therefore, it is important to conduct a study investigating systematically the potential risk factors for epilepsy.

This is a cross-sectional and hospital -based study. The participants include 80 child and adolescents who are 6 to 18 years old and 80 control subjects. The instruments include the Chinese version of Child Behavior Checklist (CBCL), 36-Item Short Form Health Survey (SF-36), Child Attitude Toward Illness Scale (CATIS), the Swanson, Nolan, and Pelham, version IV (SNAP-IV), Parental Bonding Instrument (PBI), Family APGAR, Chinese Health Questionnaire (CHQ-12), impact of childhood illness scale, drug compliance scale. We will also collect related information from chart record, and then analyze for emotion/behavior presentation and to identify the risk factors for epilepsy.

We expect that this study will reach the following objectives:

1. to understand the characteristics and prevalence of emotion/behavior problems and attention deficit hyperactivity syndrome in child and adolescents with epilepsy.
2. to investigate significant risk factors and the possible pathogenic pathway
3. to refer child and parents who have emotion problems
4. to combine research and service across departments (departments of neurology and psychiatry )
5. to improve worldwide understanding of epilepsy by the results of this study

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents had the clinical diagnosis of epilepsy
* Their ages range from 6 to 15.

Exclusion Criteria:

The subjects will be excluded from the study if they have:

* Chromosomal disorders
* Hereditary metabolic disorders
* Neurodegenerative disease
* Brain tumor; and
* Brain injury.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: clinical sample
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2007-07; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Study Director — Dept of Psychiatry, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan